CLINICAL TRIAL: NCT05725551
Title: Three Applıed Durıng Intramuscular Injectıon In Chıldren Effect Of Dıfferent Method On Paın And Fear
Brief Title: The Effect of Shotblocker, Finger Puppet And Balloon Method During Intramuscular Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Didem Lafci, Dr. Faculty Member,pHD, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MU
Record Dates: First submitted 2023-01-12; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Children

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ShotBlocker group (Experimental): Pain in intramuscular injection It is a noninvasive, plastic tool used to reduce.
  Interventions: Device: ShotBlocker
- Finger Puppet group (Experimental): Finger puppetry is an alternative method of interacting with the child through play while performing an intramuscular injection.
  Interventions: Other: Finger Puppet group
- Balloon group (Experimental): Balloon inflation method, the child inflating the balloon while performing an intramuscular injection.
  Interventions: Other: Balloon group
- Control Group (No Intervention): Intramuscular injection without any intervention.

INTERVENTIONS:
Device: ShotBlocker — Before the procedure, the protruding surface of the vehicle was placed on the injection site in contact with the skin and used by holding it during injection. The level of pain and fear experienced by the child during and 5 minutes after the injection was evaluated with the "Facial Expressions Pain Scale" and "Visual Comparison Scale", and the level of fear was evaluated with the "Child Fear Scale" by the child, the parent accompanying the child, and the observer.
  Arms: ShotBlocker group
Other: Finger Puppet group — During the interaction between the finger puppet and the child, an intramuscular injection was made. The level of pain experienced by the child during the injection and 5 minutes after the injection was evaluated by the child, the parent and the observer through the "Facial Expressions Pain Scale" and the "Visual Comparison Scale", and the fear level by the "Child Fear Scale".
  Arms: Finger Puppet group
Other: Balloon group — An intramuscular injection was given when the child began to inflate the balloon. The level of pain experienced by the child during the injection and 5 minutes after the injection was evaluated by the child, the parent and the observer through the "Facial Expressions Pain Scale" and the "Visual Comparison Scale", and the fear level by the "Child Fear Scale".
  Arms: Balloon group

SUMMARY:
The aim of the randomized controlled study is to examine the effects of ShotBlocker, finger puppet and balloon inflation methods applied during intramuscular injection procedure on children's pain and fear level.

DETAILED DESCRIPTION:
The aim of the randomized controlled study is to examine the effects of ShotBlocker, finger puppet and balloon inflation methods applied during intramuscular injection procedure on 7-12 age group children on pain and fear level.

The purpose of the research and all the working processes were explained to the children and parents by the researcher.

Children who met all eligibility criteria were invited to participate in the study with their parents.

The children and their parents were informed about the study, they were included in the study by announcing that they would be in one of the four groups, and this group was randomly determined.

Before starting the application, verbal and written consent was obtained from the parents of the children by reading/reading the Informed Voluntary Consent Form.

The child and parent were informed by the researcher about the pain and fear level assessment tools and application before and after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Children who volunteered to participate in the study and who met the inclusion criteria

Exclusion Criteria:

* Children who did not volunteer to participate in the study

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 148 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Child Fear Scale | 1 day
  The scale is a visual measurement tool consisting of five drawn facial expressions ranging from neutral expression (0=no anxiety) to frightened face (4=severe anxiety) and scores between 0-4 points.The level of pain experienced by the children in all groups during the injection and 5 minutes after the injection was evaluated.
Facial Pain Scale | 1 day
  Graded according to the severity of the pain, the leftmost face consists of "no pain" and the rightmost face consists of a total of 6 facial expressions, such as "too much pain". Faces expressing the increase in pain intensity from left to right are scored as 0,2,4,6,8,10, respectively.The level of fear experienced by the children in all groups during the injection and 5 minutes after the injection was evaluated.
Visual Analog Scale | 1 day
  The scale consists of a 10 cm / 100 mm long ruler that can be used horizontally or vertically, with "no pain" at one end and "worst pain imaginable" at the other. The child is asked to mark a spot on the line that will accurately reflect his or her pain.The level of pain experienced by the children in all groups during the injection and 5 minutes after the injection was evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Diğdem Lafcı pHD, Principal Investigator — Mersin University
Locations (1):
- Mersin University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No